CLINICAL TRIAL: NCT01057966
Title: Bioavailability of Nutrients Contained in Softgel Capsules vs Tablets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SMA-09-32
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Vision
Keywords: Bioavailability; Ocular Vitamins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ICAPS AREDS Softgel Capsule - Full Strength (Experimental): ICAPS Eye Vitamin and Mineral Supplement - Softgel
  Interventions: Dietary Supplement: ICAPS Eye Vitamin and Mineral Supplement - Softgel (full strength)
- ICAPS AREDS Softgel Capsule - Half Strength (Experimental): ICAPS Eye Vitamin and Mineral Supplement - Softgel (half -strength)
  Interventions: Dietary Supplement: ICAPS Eye Vitamin and Mineral Supplement - Softgel (half strength)
- ICAPS AREDS coated tablets - Full Strength (Experimental): ICAPS Eye Vitamin and Mineral Supplement - Coated Tablets
  Interventions: Dietary Supplement: ICAPS Eye Vitamin and Mineral Supplement - Coated Tablets (full strength)

INTERVENTIONS:
Dietary Supplement: ICAPS Eye Vitamin and Mineral Supplement - Softgel (full strength) — Single full strength dose capsule taken one time
  Arms: ICAPS AREDS Softgel Capsule - Full Strength
Dietary Supplement: ICAPS Eye Vitamin and Mineral Supplement - Softgel (half strength) — Single half strength dose capsule taken one time
  Arms: ICAPS AREDS Softgel Capsule - Half Strength
Dietary Supplement: ICAPS Eye Vitamin and Mineral Supplement - Coated Tablets (full strength) — Single, full strength dose tablet taken one time
  Arms: ICAPS AREDS coated tablets - Full Strength

SUMMARY:
This study is a comparison of the bioavailability of nutrients contained in softgel capsules vs tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 35
2. Body Mass Index (BMI) 21-27 kg/m2
3. Must be able to give written informed consent
4. Subjects must be willing to comply with all study requirements.
5. Subjects must understand, sign and be given a copy of the written Informed Consent form.

Exclusion Criteria:

1. Subjects for whom both eyes do not meet all inclusion criteria and either eye meets exclusion criteria
2. Subjects who are pregnant, lactating or planning to be pregnant during the course of the study
3. Subjects with known sensitivity to planned study concomitant medications
4. Subjects participating in any other ophthalmic drug or device clinical trial within 30 days of this clinical investigation.
5. Use of ocular drugs, other than study medications, during the study and within 14 days prior to study entry or any other ocular medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Bioavailability of nutrients | 1 week for each treatment cross-over period

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States